CLINICAL TRIAL: NCT07346638
Title: A Pilot Study of the Building Empowerment and Resilience Program for Suicidal Ideation
Brief Title: The BEAR Program for Women With Trauma Who Have Suicidal Thoughts
Acronym: BEAR-SI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Keller, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 79226
Record Dates: First submitted 2025-12-19; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Interpersonal Trauma; Depression; PTSD; Anxiety; Suicidal Ideations; Sexual Assault
Keywords: interpersonal trauma; sexual assault; suicidal ideation; self-defense
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Anxiety Disorders; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BEAR therapy group (Experimental): BEAR therapy intervention
  Interventions: Behavioral: BEAR-SI

INTERVENTIONS:
Behavioral: BEAR-SI — The BEAR Therapeutic program is a twelve-week group that meets once per week for 1.5 hours per week. The program includes three main components. The first is a psycho-educational component which provides current information about assault statistics, common risk factors, myths that are often associated assault, and safety related information The second component focuses on the development of an assortment of interpersonal skills. This part of the group offers skills such as assertiveness or communication training, boundary setting, and coping skills. The third component of our intervention consists of a thorough set of self-defense skills that help women to keep themselves safe. The repertoire of skills include recognizing unsafe situations, utilizing one's voice, and release from holds. This section provides ample practice blocks, resistance skills, and specific techniques to keep one's self safe.

SUMMARY:
The current study aims to test the feasibility of a new form of group therapy for women who have a history of interpersonal trauma and current suicidal ideation. The Building Empowerment and Resilience (BEAR) Therapeutic group has been adapted for women who have experienced trauma and have current suicidal ideation. It incorporates psychological skills, psychoeducation about trauma and gender-based violence, and physical self-defense training, all within a therapeutic process. It will be implemented with women who have experienced interpersonal trauma (physical, sexual, or emotional abuse/neglect) and experience various mental health difficulties, including suicidal ideation. We aim to assess the feasibility to recruit and implement the BEAR group. Our ultimate aim is to assess whether the program can effect self-efficacy and suicidal ideation.

DETAILED DESCRIPTION:
In the US, approximately 36% of women experience some type of sexual violence in their lifetime. Sexual violence can have a significant and lifelong impact on a women's life, with particularly high rates of mental health issues (e.g., depression, anxiety, PTSD). Women who are sexually assaulted have a three-fold risk of lifetime suicidal ideation and more than a five-fold elevated risk of suicide attempts compared to women who have not been sexually assaulted. Women who are victimized are at higher risk of subsequent sexual victimizations, and with that, worsened well-being and an even higher suicide risk.

Empowerment self-defense (ESD) training has consistently been shown to reduce the risk of both attempted and completed sexual assault by approximately 50%. Survivors of rape who participate in such training demonstrate decreases in PTSD symptoms and self-blame for past assaults. Increases in perceived self-efficacy is one of the positive outcomes of ESD work. Perceived self-efficacy is one's beliefs about their competency and capabilities to perform and is a key factor of how people think, behave, feel, and motivate themselves and how they respond in various situations, including risky or traumatic situations. Higher coping self-efficacy buffers individuals who experience trauma from posttraumatic distress, and separately, higher self-efficacy has been shown to be a protective factor against suicidality in several populations.

The purpose of the current study is to test the feasibility of the Building Empowerment and Resilience (BEAR) program which was adapted for women who have a history of sexual violence and currently endorse suicidal thinking. The Building Empowerment and Resilience-SI (BEAR-SI) Therapeutic program incorporates psychological skills, psychoeducation, and physical self-defense training, all within a therapeutic process. Our experience indicates survivors of sexual violence seek a more active intervention as they often continue to feel quite vulnerable with therapy alone. The program specifically addresses the sequalae of sexual assault and teaches skills for maintaining personal safety and for coping with unwanted thoughts, including suicidal thinking. Our goal is to determine the feasibility of the adapted BEAR program and if it enhances self-efficacy and decreases suicidal thoughts. This is a 12-week, in-person therapy group. We will examine pre- and post-group outcomes, as well as 3- and 12-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-75
* History of physical, sexual, and/or sexual emotional violence, with subsequent interpersonal or psychological distress (e.g., depression or anxiety) related to this history.
* Current suicidal thinking

Exclusion Criteria:

* Active, significant substance abuse, which could interfere with participation
* Significant medical conditions that would preclude safe participation in the study
* No history of interpersonal trauma
* Acute psychiatric instability
* History of assaultive behavior or is judged to be a potential risk to assault others.
* No current suicidal ideation or behaviors
* Unable to commit to the group for 12 weeks in-person

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Coping self-efficacy | Baseline to 12 weeks (post-group)
  This scale ranges from 0-286, with 0 indicating no confidence in managing stressors to 286 indicating very high level of confidence that one could do a particular behavior
Beck Scale for Suicidal Ideation | Baseline to 12 weeks (post-group)
  Assesses amount of suicidal thinking. The total BSS score can range from 0, with no suicidal thinking to 38 points, severe level of suicidal thinking.

OTHER OUTCOMES:
Retention in the group | 12 weeks (post-group)
  Will examine number of participants who completed at least 10/12 sessions

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keller, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study to determine the feasibility of this group. We will be collecting both qualitative and quantitative data on a small group of participants.

REFERENCES:
- [Background] Hollander, J. A., & Cunningham, J. (2020). Empowerment Self-Defense Training in a Community Population. Psychology of Women Quarterly, 44(2), 187-202. https://doi-org.laneproxy.stanford.edu/10.1177/0361684319897937
- [Background] Smith, S.G., et al. (2017). The National Intimate Partner and Sexual Violence Survey (NISVS): 2010-2012 State Report. Atlanta, GA: National Center for Injury Prevention and Control, Centers for Disease Control and Prevention.
- [Background] Denneson LM, Smolenski DJ, Bauer BW, Dobscha SK, Bush NE. The Mediating Role of Coping Self-Efficacy in Hope Box Use and Suicidal Ideation Severity. Arch Suicide Res. 2019 Apr-Jun;23(2):234-246. doi: 10.1080/13811118.2018.1456383. Epub 2018 Jul 11. PMID 29624123
- [Background] Cieslak R, Benight CC, Caden Lehman V. Coping self-efficacy mediates the effects of negative cognitions on posttraumatic distress. Behav Res Ther. 2008 Jul;46(7):788-98. doi: 10.1016/j.brat.2008.03.007. Epub 2008 Mar 18. PMID 18456241
- [Background] Dworkin ER, DeCou CR, Fitzpatrick S. Associations between sexual assault and suicidal thoughts and behavior: A meta-analysis. Psychol Trauma. 2022 Oct;14(7):1208-1211. doi: 10.1037/tra0000570. Epub 2020 Mar 23. PMID 32202845